CLINICAL TRIAL: NCT06199427
Title: Safety and Efficacy of Cyclophosphamide and Ruxolitinib for Graft-versus-host-disease Prophylaxis After Hematopoietic Stem Cell Transplantation With Thymoglobulin Serotherapy in Conditioning Regimen in Patients With Inborn Errors of Immunity
Brief Title: PTCy and and Ruxolitinib for GVHD Prophylaxis After HSCT With Thymoglobulin in Conditioning Regimen in Patients With Inborn Errors of Immunity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEI-PTCy 2023
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Inborn Errors of Immunity
MeSH Terms: interventions — Cyclophosphamide; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): Conditioning regimen containing treosulfan 30-42 g/m2, fludarabine 150 mg/mg, thymoglobulin 5 mg/kg and thiotepa 10 mg/kg or melphalan 140 mg/m2
  GVHD prophylaxis regimen for matched unrelated (MUD) and matched related donors (MRD):
  Cyclophosphamide (PTCY) 25 mg/kg/day (days +3, +4) Ruxolitinib 7 mg/m2 from day +5
  GVHD prophylaxis regimen for mismatched related donor (MMRD):
  Cyclophosphamide (PTCY) 50 mg/kg/day (days +3, +4) Ruxolitinib 7 mg/m2 from day +5
  Interventions: Drug: Cyclophosphamide; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 25mg/kg (days +3, +4) after HSCT from MUD and MRD Cyclophosphamide 50mg/kg (days +3, +4) after HSCT from MMRD
Drug: Ruxolitinib — Ruxolitinib 7 mg/m2 from day +5 after HSCT

SUMMARY:
The aim of the current study is to evaluate the efficacy of combined regimen of GVHD prophylaxis with thymoglobulin in conditioning regimen and PTCY with ruxolitinib used after HSCT in patients with inborn errors of immunity (IEI)

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is widely used in inborn errors of immunity (IEI), and risks of graft-versus-host disease (GVHD) remain high. Use of post-transplant cyclophosphamide (PTCY) for GVHD prophylaxis revolutionized the outcomes of HSCT from mismatched related donor (MMRD). Use of ruxolitinib for GVHD prophylaxis demonstrates promising results in adult patients. Another well-known option for GVHD prevention is antithymocyte globulin. To evaluate the efficacy of combination of thymoglobulin with PTCY and ruxolitinib for GVHD prophylaxis, conditioning regimen containing treosulfan 30-42 g/m2, fludarabine 150 mg/mg, and thiotepa 10 mg/kg or melphalan 140 mg/m2 and GVHD prophylaxis regimen containing cyclophosphamide 50 mg/kg for MMRD, 25 mg/kg for matched unrelated and related donors at days +3, 4 post-HSCT and ruxolitinib at dose 7 mg/m2 from day +5 after HSCT will be used in patients with IEI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 0 months and < 21 years
2. Patients diagnosed with NBS eligible for an allogeneic HSCT
3. Signed written informed consent signed by a parent or legal guardian

Exclusion Criteria:

Concomitant severe somatic disease associated with an additional risk of severe complications

Ages: 0 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 1 year after HSCT
  Events: graft failure, death

SECONDARY OUTCOMES:
Overall survival | 1 year after HSCT
Cumulative incidence of acute graft versus host disease | 1 year after HSCT
Cumulative incidence of chronic graft versus host disease | 1 year after HSCT
Cumulative incidence of engraftment | 100 days
Cumulative incidence of graft failure | 1 year after HSCT
Incidence of early organ toxicity | 100 days
Cumulative incidence of transplant related mortality | 1 year after HSCT
Cumulative incidence of viral infections | 1 year after HSCT
Investigation of the concentration of ruxolitinib in the blood To investigate the pharmacokinetics of ruxolitinib | 1 month after HSCT
  The features of pharmacokinetics in children of different ages

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Balashov, MD, PhD, Study Chair — National Research Center for Pediatric Hematology, Moscow, Russia
Locations (1):
- HSCT department, Moscow, Russia